CLINICAL TRIAL: NCT00862888
Title: A 2-Cohort, Multi-Centre, Randomised, Double Blind, Placebo Controlled 4-Way Crossover Study To Assess The Efficacy Of Single Oral Doses Of PF-00446687 On Erectile Function In Men Suffering From Erectile Dysfunction, Using 100 Mg Sildenafil As A Positive Control.
Brief Title: Study to Investigate Effect of a New Drug (PF-00446687) in Males Suffering From Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A8361011
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — 1-((1-tert-butyl-4-(2,4-difluorophenyl)pyrrolidin-3-yl)carbonyl)-3,5-dimethyl-4-phenylpiperidin-4-ol; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1; Study Period 1, 2, 3 or 4 (Placebo Comparator): Cohort 1: Exploring two single doses of PF-00446687 200 mg as well as sildenafil 100mg and placebo (double dummy design)
  Interventions: Drug: PF-00446687; Drug: Placebo; Drug: Sildenafil
- Cohort 2; study periods 1, 2, 3 or 4 (Placebo Comparator): Cohort 2: Exploring single doses of PF-00446687 20 mg - 175 mg. Subjects to receive two of 3 possible doses of PF-00446687 as well as a single dose of sildenafil 100mg and placebo (double dummy design).
  Interventions: Drug: PF-00446687; Drug: Placebo; Drug: Sildenafil

INTERVENTIONS:
Drug: PF-00446687 — Single 200mg dose as an oral solution
  Arms: Cohort 1; Study Period 1, 2, 3 or 4
Drug: Placebo — Placebo for oral solution
  Arms: Cohort 1; Study Period 1, 2, 3 or 4
Drug: Placebo — Placebo for tablet
  Arms: Cohort 1; Study Period 1, 2, 3 or 4
Drug: Sildenafil — Single oral dose 100 mg tablet
  Arms: Cohort 1; Study Period 1, 2, 3 or 4
Drug: PF-00446687 — Single 125 mg dose as an oral solution
  Arms: Cohort 2; study periods 1, 2, 3 or 4
Drug: PF-00446687 — Single 175 mg dose as an oral solution
  Arms: Cohort 2; study periods 1, 2, 3 or 4
Drug: PF-00446687 — Single 20 mg dose as an oral solution
  Arms: Cohort 2; study periods 1, 2, 3 or 4
Drug: Placebo — Placebo for oral solution
  Arms: Cohort 2; study periods 1, 2, 3 or 4
Drug: Placebo — Placebo for tablet
  Arms: Cohort 2; study periods 1, 2, 3 or 4
Drug: Sildenafil — Single oral dose 100 mg tablet
  Arms: Cohort 2; study periods 1, 2, 3 or 4

SUMMARY:
The purpose of this study is to investigate the effect of up to 200 mg of PF-00446687 on erectile activity in males suffering from erectile dysfunction as well as examining the safety and toleration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-65 years who has given written informed consent to participate in the study and who suffers moderate to severe erectile dysfunction who has a current or recent successful response to treatment with phosphodiesterase type 5 inhibitors

Exclusion Criteria:

* Males with a history of significant cardiac disease; unstable angina or recent myocardial infarction.
* Males suffering from treated or untreated hypo- or hypertension
* Males currently receiving vasoactive medication
* Males taking medications contraindicated, or cautioned with sildenafil or MC4 agonists

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Assess effect of single doses of PF-00446687 on erectile function (using the Rigiscan+ device) | Day of dosing
Evaluate subjective self-assessment of sexual interest and desire by means of a questionnaire | Day of dosing
Diary of sexual activities | From day of dosing to 7 days post-dose

SECONDARY OUTCOMES:
PK assessment of PF-00446687 ad sildenafil | Day of dosing
Safety and toleration | Day of dosing to follow-up
Assess variability of response and repeatability of design between 2 similar doses | Comparison of response to be assessed until 7 days post-dose
Assess agouti related protein levels in this population | Day of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Oslo, Norway
- United Kingdom (2):
  - Pfizer Investigational Site, Belfast, Northern Ireland
  - Pfizer Investigational Site, Leeds, WEST Yorkshire

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8361011&StudyName=Study%20to%20investigate%20effect%20of%20a%20new%20drug%20%28PF-00446687%29%20in%20males%20suffering%20from%20erectile%20dysfunction